CLINICAL TRIAL: NCT03878641
Title: Literacy and Language Interventions Via Telepractice for School-Age Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Shih-Yuan Liang, Principal Investigator, Vanderbilt University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Telepractice
Record Dates: First submitted 2019-03-15; First posted 2019-03-18 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Literacy-language Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Children in Grade 1 to 5 with literacy and language needs (Experimental): The investigators intend to identify children in Grade 1 to 5 who demonstrate language-based learning difficulties. Using the two-stage screening, the investigators will identify children who produce substantial number of reading miscues and/or self-correct more less 25% of their miscues, and/or who present weaknesses in expressive language skills with a total CUBED score lower than grade-specific cut scores.
  Interventions: Behavioral: Children in Grade 1 to 5 with literacy and language needs

INTERVENTIONS:
Behavioral: Children in Grade 1 to 5 with literacy and language needs — The investigators deliver a telepractice-based intervention targeting: (a) Word reading and phonics instruction, (b) applying a comprehension monitoring strategy to improve text reading accuracy, and (c) complex sentences use in written text. Participants receive 3 online 50-minute tutoring session weekly across 15 weeks.

SUMMARY:
Telepractice refers to the application of telecommunication technology (e.g., Skype, Webex, Zoom) to the delivery of speech-language and audiology services. The development of telepractice, an emerging alternative to traditional service delivery, has been driven by the need for equitable access and cost-effective services to all client, regardless of geographical locations, physical conditions, or social and economic status (Theodoros, 2011).

The purpose of this study is to examine the feasibility of telepractice-delivered intervention targeting literacy (i.e., reading and writing) and literate language skills (e.g., narrative skills) to promote better academic outcomes in school-age children. The investigators conduct a single-subject, multiple probe design across four participants to examine the functional relation between a telepractice intervention and two educational outcomes - reading self-corrections and narrative ability. Participants with language and literacy needs receive three weekly intervention sessions via ZOOM (a videoconferencing software). A single-subject, multiple-probe design across participants enables the examination of treatment effectiveness: If three replications of treatment effect are established across participants (i.e., visual analysis indicates evident behavioral change on progress-monitoring assessment), the proposed intervention yields a high likelihood of producing benefits to children who share similar learning needs.

In addition to intervention effectiveness of telepractice, the investigators examine feasibility along two dimensions: Fidelity and scoring reliability. Fidelity here includes two components - fidelity of intervention (i.e., whether the intervention activities are implemented as intended) and procedural fidelity of probe assessment administration (whether the progress-monitoring probes are administered as intended). Scoring reliability (e.g., interobserver agreement) examines if the interventionist's scoring is consistent with a reliability coder's scoring. Evidence derived from analyses of fidelity, reliability, and intervention effectiveness will be examined collectively to determine the feasibility of delivering literacy and language intervention via telepractice.

DETAILED DESCRIPTION:
The single-subject multiple-probe design comprises four phases: (a) eligibility determination, (b) a baseline condition, wherein participants receive business-as-usual practice, (c) a 15-week intervention condition, and (d) a maintenance condition (see Figure 1).

Eligibility determination. The investigators employ a two-stage screening procedure (psycho-educational assessments) to identify children in Grade 1 to 5 who demonstrate language-based learning difficulties. Following the completion of the two-stage screening, the investigators conduct a mock tutoring session to familiarize the potential participants with the technology platform. The interventionist fills out a behavior checklist that consists of steps needed to be accomplished in the mock session to determine if the child meets the minimum criteria for telepractice candidacy.

Baseline condition. In the baseline condition, the interventionist meets with each participant three times a week to collect baseline data. Participants receive business-as-usual instruction-that is, the interventionist stops the child immediately at point of miscues, supplies the word, and tells the child to continue reading.

Intervention condition. The proposed intervention program consists of three components: (a) Word reading and phonics instruction, (b) applying a comprehension monitoring strategy to improve text reading accuracy, and (c) complex sentences use in written text. With each participant, instruction is delivered in three 50-minute weekly sessions across 15 weeks. Intervention activities delivered in the first, second, and third session of the week is outlined in Figure 1. The interventionist collects the CUBED Narrative Language Measure (NLM) probe on the fourth day of the week when no instruction is given. The 3-minute reading probes will be administered on a weekly basis.

Maintenance condition. Across three weeks of no intervention, each of the progress-monitoring assessments is administered once per week.

ELIGIBILITY:
Inclusion Criteria:

* Children who produce substantial number of reading miscues and/or self-correct more less 25% of their miscues, and/or who present weaknesses in expressive language skills with a total CUBED score lower than grade-specific cut scores.

Exclusion Criteria:

* Additional exclusionary criteria include: (a) nonverbal IQ standard score > 80 and (b) no reported history of autism, hearing loss, visual impairment, or other neurological disorder (c) meet the criteria for telepratice candidacy (as informed by a behavior checklist filled out by the examiner).

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2019-04-29 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Reading Comprehension | Baseline to 4 months
  The Passage Comprehension subtest of the Woodcock Reading Mastery Test-3rd edition (WRMT-III) and the Reading Comprehension test of the Wechsler Individual Achievement Test-3rd edition (WIAT-III) will be administered to assess a child's reading comprehension

SECONDARY OUTCOMES:
Complex sentence use in narrative production | Weekly for 4 months
  The investigators count the instances of dependent clauses and T-units (operationalized as an independent clause plus its dependent clause[s]). We divide the number of dependent clause tokens by the number of T-units to form the index of complex sentence proportion.
Reading self-correction in independent oral reading | Weekly to 4 months
  The Curriculum-Based Measurement Passage Reading Fluency probe is administered twice weekly to monitor a child's progress in self-correction proportion. The primary dependent variable, self-correction proportion, is operationalized as the number of self-corrections divided by the number of reading miscues produced in a 3-minute reading probe.

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Schuele, PhD, Study Chair — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No